CLINICAL TRIAL: NCT05424432
Title: Short Course Neoadjuvant Chemo-radiotherapy Plus Anti-PD-1 Antibody (Toripalimab) for Locally Advanced Resectble Squamous Cell Carcinoma of Esophagus (SCALE-2）
Brief Title: Short Course Neoadjuvant Chemo-radiotherapy Plus Toripalimab for Locally Advanced Resectble Squamous Cell Carcinoma of Esophagus
Acronym: SCALE-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Ning Jiang, M.D./Ph.D., M.D., Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCALE-2
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Locally Advanced Esophageal Carcinoma
Keywords: esophageal carcinoma; short course neoadjuvant radiotherapy; Toripalimab; neoadjuvant chemoradiotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- short course neoadjuvant chemoradiotherapy plus toripalimab (Experimental): Paclitaxel, carboplatin and toripalimab every 3 weeks for two cycles. Concurrent short course neoadjuvant radiotherapy (30 Gy in 12 fractions, 5 days per week, D3-D18).
  Surgery will be performed within 8-10 weeks after the completion of preoperative therapy described above.
  Interventions: Drug: Neoadjuvant Chemotherapy; Drug: Neoadjuvant Toripalimab; Radiation: Short Course Neoadjuvant Radiotherapy

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy — Paclitaxel (135 mg /m2) and carboplatin (AUC=5) every 3 weeks for two cycles (D1,D22)
Drug: Neoadjuvant Toripalimab — Toripalimab 240mg every 3 weeks for two cycles (D2,D23)
Radiation: Short Course Neoadjuvant Radiotherapy — 30 Gy in 12 fractions, 1 fraction per day, 5 days per week, D3-D18

SUMMARY:
Adding PD-1 inhibitors to neoadjuvant chemoradiotherapy has shown promising results in locally advanced resectable esophageal squamous cell carcinoma (ESCC). However, there is a need to explore safer and more effective treatment doses and schedules. This is an open labeled, prospective, single-arm phase II trial to evaluate the safety and efficacy of the short course neoadjuvant chemo-radiotherapy plus Toripalimab for locally advanced resectble ESCC.

DETAILED DESCRIPTION:
Although neoadjuvant chemoradiotherapy (CRT) followed by surgery has become the standard treatment option for locally advanced ESCC, prognosis of these patients is still poor. Adding PD-1/PD-L1 checkpoints inhibitor to neoadjuvant chemoradiotherapy (CRT) have shown potential benefit in locally advanced resectble ESCC. However, the conventional radiation dose may lead to irreversible toxicity. There is need to explore more effective and safer treatment doses and schedules for this combination.

The investigators proposed a novel strategy (short course neoadjuvant radiotherapy plus preoperative chemotherapy and toripalimab, the SCALE strategy) for the treatment of locally advanced resectble ESCC. In the phase Ib SCALE-1 (ChCTR2100045104) study, 23 patients were enrolled and 20 patients had undergone surgery after the preoperative treatment. The preliminary results showed that the SCALE strategy was safe and induced a pCR and MPR in 55% and 80% of resected tumors, respectively. In this prospective, phase II study, the investigators will further evaluate the safety and efficacy of the SCALE strategy in locally advanced resectble ESCC. This study will provide valuable information for further clinical use of SCALE strategy in locally advanced resectble ESCC.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to provide written informed consent and understand and agree to follow the research requirements and evaluation schedule.
2. Endoscopic biopsy of thoracic esophageal primary lesion histologically diagnosed as squamous cell carcinoma.
3. Clinical stage T1-4aN+M0 or T3-4aN0M0 in the UICC-TNM classification 8th edition.
4. The age is over 20 years old and under 75 on the enrollment date (including 20 and 75), including both female and male.
5. PS 0-1.
6. According to RECIST version 1.1, there were measurable or evaluable lesions.
7. No medical history of treatment for cancer (No medical history of chemotherapy, radiotherapy and endocrine therapy, immune-therapy or other study drugs including treatment for other types of cancer).
8. The results of laboratory tests within 14 days before enrollment meet the inclusion criteria：（patients should not receive blood transfusion or growth factor support because neutrophil count, platelet or hemoglobin are lower than the research requirements within 14 days before blood sample collection）.

   * Bone marrow function: hemoglobin (Hb) >=90g/L; white blood cell count (WBC) >= lower limit of normal value; absolute neutrophil value (ANC) >= 1.5x10^9 /L; platelet count >= 100x10^9 / L;
   * Renal function: Cr <= 1.5 UNL, endogenous creatinine clearance rate (Ccr) >= 60 ml/min（Cockcroft-Gault）;
   * Liver function: total bilirubin <= 1.5 ULN; ALT and AST <= 2.5 ULN (patients with liver metastases can be relaxed to <=5 ULN);
   * Blood coagulation function: the international standardized ratio of prothrombin time <= 1.5 ULN, and the partial thromboplastin time is within the normal range.
9. Patients with hepatitis B virus (HBV) infection, inactive / asymptomatic HBV carriers, or patients with chronic or active HBV will be allowed to be enrolled if HBV DNA < 500 IU / ml (or 2500 copies / ml) at screening. Patients with positive hepatitis C antibody will be allowed to be enrolled if HCV-RNA is negative during screening.Note: patients who can detect hepatitis B surface antigen (HBsAg) or HBV DNA should be treated with antiviral drugs for more than 2 weeks before enrollment, and the treatment should be continued for 6 months after the study drug treatment.
10. Women of childbearing age (wocbp) should take the urine or serum pregnancy test, and the result of which should be negtive within ≤ 72 hours before treatment. For females, who have agreed with contraception from start of investigational drug administration to 5 months after last dose of investigational drug. For males who have agreed with contraception from start of investigational drug administration to 7 months after last dose of investigational drug.

Exclusion Criteria:

1. Have received any treatment for esophageal squamous cell carcinoma in the past;
2. Patients with evidence or high risk of gastrointestinal hemorrhage or fistula (esophagus / bronchus or esophagus / aorta);
3. Patients with severe malnutrition, with body mass index lower than 18.5kg/m2, or PG-SGA score ≥9；
4. Any active autoimmune disease or history of autoimmune disease (as follows, but not limited to: interstitial pneumonia, uveitis, enteritis, autoimmune hepatitis, pituitritis, vasculitis, nephritis, hyperthyroidism, thyroid dysfunction); Subjects with vitiligo or who have had complete remission from childhood asthma without any intervention after adulthood may be included; Asthma requiring medical intervention with bronchodilators was not included.
5. Has a previous radiotherapy, chemotherapy, hormone therapy, surgery, molecular targeted therapy or immune therapy for this malignancy or for any other past malignancy;
6. Any condition requiring systemic corticosteroid therapy (prednisone with a dose higher than 10 mg / day or equivalent dose of similar drugs) or other immunosuppressants within 14 days before treatment. （Excluding the following steroid regimens：Local, ophthalmic, intra-articular, nasal and inhaled corticosteroids with minimal systemic absorption；Prophylactic short-term (≤ 7 days) use of corticosteroids (e.g., prevention of contrast media allergy) or for the treatment of non-autoimmune disorders (e.g., delayed hypersensitivity caused by exposure to allergens).
7. Live vaccine injection was received in ≤ 4 weeks before treatment.
8. A history of immunodeficiency, including HIV infection, other acquired or congenital immunodeficiency, or a history of organ or bone marrow implantation that need immunosuppressive medications.
9. There are clinical symptoms or diseases of the heart that are not well controlled, such as: 1). heart failure above grade 2 by the Criteria of NYHA; 2). unstable angina pectoris; 3). myocardial infarction occurred within 1 year; 4). Clinically meaningful supraventricular or ventricular arrhythmias require treatment or intervention;
10. Has severe infections （CTCAE>2 grade）within 4 weeks before treatment; basal thoracic imaging indicating active pneumonia, or other infectious situation that need oral or intravenous antibiotic treatment (excluding Prophylactic medication for antibiotics).
11. A history of interstitial lung disease, non-infectious pneumonia or uncontrolled disease, including pulmonary fibrosis, acute lung disease, etc.
12. Has active pulmonary tuberculosis found by CT imaging; or has active pulmonary tuberculosis less than 1 year before inclusion; or has active pulmonary tuberculosis but without standard treatment over 1 year before inclusion;
13. Allergic to any drug used in this study.
14. Pregnant or lactating women；participants who unwilling to take contraception.
15. Other factors that could lead to the termination of this study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | 1 month after resection
  Pathologic complete response was defined as pT0N0M0 or pTisN0M0

SECONDARY OUTCOMES:
Disease free survival | 3 years after resection
  Disease free survival defined as the time from enrollment to the first documented disease progression of local recurrence or distant metastasis or death due to any cause.
3-year overall survival | 3 years after enrollment
  Defined as from date of enrollment until the date of death from any cause or the date of last follow-up, whichever came first.
Incidence of Treatment-related Adverse Events | From the date of enrollment until surgery was applied during study period or up to at least 90 days after last dose
  The neoadjuvant treatment-related adverse events as assessed by CTCAE v5.0
Perioperative complication rate | From date of surgery to 30 days later
  The perioperative complication rate of esophagectomy using clavien-Dindo classification
Health related quality of Life | Measured before and after neoadjuvant therapy, before and 1, 3, 6, 9, 12 months after surgery.
  To compare change in Quality of Life, as defined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30 (Version 3)) during the neoadjuvant therapy and perioperative period.
  The EORTC QLQ-C30 (Version 3) uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
  The EORTC QLQ-C30 (Version 3) uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.
Health related quality of Life related to esophageal carcinoma | Measured before and after neoadjuvant therapy, before and 1, 3, 6, 9, 12 months after surgery.
  To compare change in Quality of Life in esophageal carcinoma patients, the European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire for Esophageal Cancer (EORTC QLQ-QES18) was used.
  The EORTC QLQ-QES18 uses for the questions 1 to 18 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangzhi Zhu, M.D., Study Director — Jiangsu Cancer Institute & Hospital; Ming Jiang, M.D., Study Director — Jiangsu Cancer Institute & Hospital; Feng Jiang, M.D., Study Director — Jiangsu Cancer Institute & Hospital
Locations (1):
- Jiangsu Cancer Hospital /Jiangsu Institute of Cancer Research, Nanjing, Jiangsu, China